CLINICAL TRIAL: NCT02636413
Title: Evaluation of the Impact of LacTEST on Diagnostic Thinking and on Patient Management, and of the Reproducibility (Test-Retest), for the Diagnosis of Hypolactasia in Adults and Elderly Patients Presenting With Clinical Symptoms of Lactose Intolerance
Brief Title: Evaluation of LacTEST for the Diagnosis of Hypolactasia in Adults and Elderly Patients Presenting With Clinical Symptoms of Lactose Intolerance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VenterPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VPH-GXL-2013-01; 2015-001181-26 (EudraCT Number)
Record Dates: First submitted 2015-12-10; First posted 2015-12-21 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance | interventions — 4-O-galactopyranosylxylose; Lactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LacTEST (Experimental): 0,45 g of gaxilose po, once, per diagnostic test performed.
  Interventions: Drug: gaxilose
- Hydrogen Breath Test (Active Comparator): 25 to 50 g of lactose po, once, per diagnostic test performed.
  Interventions: Dietary Supplement: lactose

INTERVENTIONS:
Drug: gaxilose — After gaxilose administration, urine collection, cuantification (firstly from 0 to 4 hours, and total urine from 0 to 5 hours), and xilose cuantification afterwards.
  Other Names: LacTEST
  Arms: LacTEST
Dietary Supplement: lactose — After lactose administration, expired hydrogen measurement at pre-specified intervals.
  Other Names: Hydrogen Breath Test (HBT)
  Arms: Hydrogen Breath Test

SUMMARY:
The purpose of this study is to evaluate both the impact of LacTEST on diagnostic thinking and on patient management, and its reproducibility (Test-Retest), for the diagnosis of hypolactasia in adults and elderly patients presenting with clinical symptoms of lactose intolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of either sex, between 18 and 70 years old.
2. Capacity for understanding and giving the informed consent to participate in this study.
3. Patients with clinical suggestive of lactose intolerance, primary or secondary, who have not been diagnosed and that fulfil the requirements allowed by the gaxilose summary of product characteristics (SmPC).

Exclusion Criteria:

1. Pregnant women or breast-feeding women.
2. Unable or reticent to give the informed consent or to comply with the study requirements.
3. Patients with glomerular filtration rate (GFR) less than 90 ml/min/1.73m2.
4. Portal hypertension: ascites, cirrhosis.
5. Medical records of total gastrectomy and/or vagotomy.
6. Patients diagnosed with myxedema.
7. Patients with Diabetes Mellitus.
8. Patients who are participating or have participated in any clinical trial within the 3 months previous to their inclusion in the study.
9. Patients who are drug abuse consumers.
10. Patients under treatment with antibiotics, sulphamides and antiparasitics, who cannot suspend the treatments 7 days prior to the performance of the hydrogen breath test.
11. Patients with any recognized and already existing disorder that might interfere with the any of the lactose intolerance diagnosis tests.
12. Patients who have taken aspirin of indomethacin in the 48h preceding the performance of the Gaxilose test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogical Scale | Through study completion, up to 10 months.
  The primary objective is to demonstrate non-inferiority of gaxilose test, compared with Hydrogen Breath Test (HBT) using a validated method (VAS results pre and post-test), on the impact on diagnostic thinking for the diagnosis of hypolactasia.

SECONDARY OUTCOMES:
Physician's Questionnaire | Through study completion, up to 10 months.
  To demonstrate non-inferiority of gaxilose test, compared with Hydrogen Breath Test (HBT), on the impact on patient management for the diagnosis of hypolactasia, through a Physician's Qestionnaire.
Intraclass Correlation Coefficient | Through study completion, up to 10 months.
  To demonstrate gaxilose test reproducibility [ICC (2,1)] with urine accumulated from 0-4h after gaxilose administration, and with urine accumulated from 0-5h after gaxilose administration.
Number of participants with treatment-related adverse events as assessed by the most recent version of MedDRA thesaurus. | Through study completion, up to 10 months.
  To assess the safety profile of both tests performed, by assessing the frecuency of treatment-related AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Crespo, MD, PhD, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (6):
- Spain (6):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Doctor Josep Trueta, Girona, Girona
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aragon JJ, Hermida C, Martinez-Costa OH, Sanchez V, Martin I, Sanchez JJ, Codoceo R, Cano JM, Cano A, Crespo L, Torres Y, Garcia FJ, Fernandez-Mayoralas A, Solera J, Martinez P. Noninvasive diagnosis of hypolactasia with 4-Galactosylxylose (Gaxilose): a multicentre, open-label, phase IIB-III nonrandomized trial. J Clin Gastroenterol. 2014 Jan;48(1):29-36. doi: 10.1097/MCG.0b013e318297fb10. PMID 23722657
- [Background] Chinn S. Statistics in respiratory medicine. 2. Repeatability and method comparison. Thorax. 1991 Jun;46(6):454-6. doi: 10.1136/thx.46.6.454. No abstract available. PMID 1858087
- [Background] Landis JR, Koch GG. An application of hierarchical kappa-type statistics in the assessment of majority agreement among multiple observers. Biometrics. 1977 Jun;33(2):363-74. No abstract available. PMID 884196
- [Background] Sahi T. Genetics and epidemiology of adult-type hypolactasia. Scand J Gastroenterol Suppl. 1994;202:7-20. doi: 10.3109/00365529409091740. PMID 8042019
- [Background] Villako K, Maaroos H. Clinical picture of hypolactasia and lactose intolerance. Scand J Gastroenterol Suppl. 1994;202:36-54. doi: 10.3109/00365529409091743. PMID 8042017
- [Background] Suchy FJ, Brannon PM, Carpenter TO, Fernandez JR, Gilsanz V, Gould JB, Hall K, Hui SL, Lupton J, Mennella J, Miller NJ, Osganian SK, Sellmeyer DE, Wolf MA. NIH consensus development conference statement: Lactose intolerance and health. NIH Consens State Sci Statements. 2010 Feb 24;27(2):1-27. PMID 20186234
- [Background] Newcomer AD, McGill DB, Thomas PJ, Hofmann AF. Prospective comparison of indirect methods for detecting lactase deficiency. N Engl J Med. 1975 Dec 11;293(24):1232-6. doi: 10.1056/NEJM197512112932405. PMID 1186802
- [Background] Jellema P, Schellevis FG, van der Windt DA, Kneepkens CM, van der Horst HE. Lactose malabsorption and intolerance: a systematic review on the diagnostic value of gastrointestinal symptoms and self-reported milk intolerance. QJM. 2010 Aug;103(8):555-72. doi: 10.1093/qjmed/hcq082. Epub 2010 Jun 3. PMID 20522486
- [Background] Shaukat A, Levitt MD, Taylor BC, MacDonald R, Shamliyan TA, Kane RL, Wilt TJ. Systematic review: effective management strategies for lactose intolerance. Ann Intern Med. 2010 Jun 15;152(12):797-803. doi: 10.7326/0003-4819-152-12-201006150-00241. Epub 2010 Apr 19. PMID 20404262
- [Background] Newcomer AD, McGill DB. Distribution of disaccharidase activity in the small bowel of normal and lactase-deficient subjects. Gastroenterology. 1966 Oct;51(4):481-8. No abstract available. PMID 5922947
- [Background] Hovde O, Farup PG. A comparison of diagnostic tests for lactose malabsorption--which one is the best? BMC Gastroenterol. 2009 Oct 31;9:82. doi: 10.1186/1471-230X-9-82. PMID 19878587
- [Background] Arola H. Diagnosis of hypolactasia and lactose malabsorption. Scand J Gastroenterol Suppl. 1994;202:26-35. doi: 10.3109/00365529409091742. PMID 8042016
- [Background] Aragon JJ, Canada FJ, Fernandez-Mayoralas A, Lopez R, Martin-Lomas M, Villanueva D. A direct enzymatic synthesis of beta-D-galactopyranosyl-D-xylopyranosides and their use to evaluate rat intestinal lactase activity in vivo. Carbohydr Res. 1996 Sep 2;290(2):209-16. doi: 10.1016/0008-6215(96)00113-9. PMID 8823908
- [Background] Hermida C, Corrales G, Canada FJ, Aragon JJ, Fernandez-Mayoralas A. Optimizing the enzymatic synthesis of beta-D-galactopyranosyl-D-xyloses for their use in the evaluation of lactase activity in vivo. Bioorg Med Chem. 2007 Jul 15;15(14):4836-40. doi: 10.1016/j.bmc.2007.04.067. Epub 2007 May 6. PMID 17512743
- [Background] Hermida C, Guerra P, Martinez-Costa OH, Sanchez V, Sanchez JJ, Solera J, Fernandez-Mayoralas A, Codoceo R, Frias J, Aragon JJ. Phase I and phase IB clinical trials for the noninvasive evaluation of intestinal lactase with 4-galactosylxylose (gaxilose). J Clin Gastroenterol. 2013 Jul;47(6):501-8. doi: 10.1097/MCG.0b013e318272f507. PMID 23328304
- [Background] Lord SJ, Irwig L, Simes RJ. When is measuring sensitivity and specificity sufficient to evaluate a diagnostic test, and when do we need randomized trials? Ann Intern Med. 2006 Jun 6;144(11):850-5. doi: 10.7326/0003-4819-144-11-200606060-00011. PMID 16754927
- [Background] Fryback DG, Thornbury JR. The efficacy of diagnostic imaging. Med Decis Making. 1991 Apr-Jun;11(2):88-94. doi: 10.1177/0272989X9101100203. PMID 1907710
- [Background] Lijmer JG, Leeflang M, Bossuyt PM. Proposals for a phased evaluation of medical tests. Med Decis Making. 2009 Sep-Oct;29(5):E13-21. doi: 10.1177/0272989X09336144. Epub 2009 Jul 15. PMID 19605881
- [Background] Van den Bruel A, Cleemput I, Aertgeerts B, Ramaekers D, Buntinx F. The evaluation of diagnostic tests: evidence on technical and diagnostic accuracy, impact on patient outcome and cost-effectiveness is needed. J Clin Epidemiol. 2007 Nov;60(11):1116-22. doi: 10.1016/j.jclinepi.2007.03.015. Epub 2007 Aug 29. PMID 17938052
- [Background] Blanchard TK, Mackenzie R, Bearcroft PW, Sinnatamby R, Gray A, Lomas DJ, Constant CR, Dixon AK. Magnetic resonance imaging of the shoulder: assessment of effectiveness. Clin Radiol. 1997 May;52(5):363-8. doi: 10.1016/s0009-9260(97)80131-6. PMID 9171790
- [Background] Stanko LK, Jacobsohn E, Tam JW, De Wet CJ, Avidan M. Transthoracic echocardiography: impact on diagnosis and management in tertiary care intensive care units. Anaesth Intensive Care. 2005 Aug;33(4):492-6. doi: 10.1177/0310057X0503300411. PMID 16119491
- [Background] Blaivas M, Kuhn W, Reynolds B, Brannam L. Change in differential diagnosis and patient management with the use of portable ultrasound in a remote setting. Wilderness Environ Med. 2005 Spring;16(1):38-41. doi: 10.1580/1080-6032(2005)16[38:ciddap]2.0.co;2. PMID 15813146
- [Background] Hobby JL, Dixon AK, Bearcroft PW, Tom BD, Lomas DJ, Rushton N, Matthewson MH. MR imaging of the wrist: effect on clinical diagnosis and patient care. Radiology. 2001 Sep;220(3):589-93. doi: 10.1148/radiol.2203001429. PMID 11526253
- [Background] Wilt TJ, Shaukat A, Shamliyan T, Taylor BC, MacDonald R, Tacklind J, Rutks I, Schwarzenberg SJ, Kane RL, Levitt M. Lactose intolerance and health. Evid Rep Technol Assess (Full Rep). 2010 Feb;(192):1-410. PMID 20629478
- [Background] Srinivasan U, Jones E, Weir DG, Feighery C. Lactase enzyme, detected immunohistochemically, is lost in active celiac disease, but unaffected by oats challenge. Am J Gastroenterol. 1999 Oct;94(10):2936-41. doi: 10.1111/j.1572-0241.1999.01441.x. PMID 10520848
- [Background] Phillips AD, Avigad S, Sacks J, Rice SJ, France NE, Walker-Smith JA. Microvillous surface area in secondary disaccharidase deficiency. Gut. 1980 Jan;21(1):44-8. doi: 10.1136/gut.21.1.44. PMID 7364319
- [Background] Kaufman SS, Lyden ER, Brown CR, Iverson AK, Davis CK, Sudan DL, Fox IJ, Horslen SP, Shaw BW Jr, Langnas AN. Disaccharidase activities and fat assimilation in pediatric patients after intestinal transplantation. Transplantation. 2000 Feb 15;69(3):362-5. doi: 10.1097/00007890-200002150-00009. PMID 10706043
- [Background] Kirschner BS, DeFavaro MV, Jensen W. Lactose malabsorption in children and adolescents with inflammatory bowel disease. Gastroenterology. 1981 Nov;81(5):829-32. PMID 6895202
- [Background] Van Biervliet S, Eggermont E, Carchon H, Veereman G, Deboeck K. Small intestinal brush border enzymes in cystic fibrosis. Acta Gastroenterol Belg. 1999 Jul-Sep;62(3):267-71. PMID 10547891
- [Background] Parnes HL, Fung E, Schiffer CA. Chemotherapy-induced lactose intolerance in adults. Cancer. 1994 Sep 1;74(5):1629-33. doi: 10.1002/1097-0142(19940901)74:53.0.co;2-l. PMID 8062196
- [Background] Bond JH, Levitt MD. Quantitative measurement of lactose absorption. Gastroenterology. 1976 Jun;70(6):1058-62. PMID 1269865
- [Background] Maxwell C. Sensitivity and accuracy of the visual analogue scale: a psycho-physical classroom experiment. Br J Clin Pharmacol. 1978 Jul;6(1):15-24. doi: 10.1111/j.1365-2125.1978.tb01676.x. PMID 666944
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Background] Hobby JL, Tom BD, Todd C, Bearcroft PW, Dixon AK. Communication of doubt and certainty in radiological reports. Br J Radiol. 2000 Sep;73(873):999-1001. doi: 10.1259/bjr.73.873.11064655.
- [Background] Dixon AK. The impact of medical imaging on the physician's diagnostic and therapeutic thinking. Eur Radiol. 1998;8(3):488-90. doi: 10.1007/s003300050423. No abstract available. PMID 9510594
- [Background] Mackenzie R, Dixon AK, Keene GS, Hollingworth W, Lomas DJ, Villar RN. Magnetic resonance imaging of the knee: assessment of effectiveness. Clin Radiol. 1996 Apr;51(4):245-50. doi: 10.1016/s0009-9260(96)80340-0. PMID 8617035
- [Background] Pitkanen E. The conversion of D-xylose into D-threitol in patients without liver disease and in patients with portal liver cirrhosis. Clin Chim Acta. 1977 Oct 1;80(1):49-54. doi: 10.1016/0009-8981(77)90262-5. PMID 908147
- [Background] CRANE RK. Intestinal absorption of sugars. Physiol Rev. 1960 Oct;40:789-825. doi: 10.1152/physrev.1960.40.4.789. No abstract available. PMID 13696269
- [Derived] Monsalve-Hernando C, Crespo L, Ferreiro B, Martin V, Aldeguer X, Opio V, Fernandez-Gil PL, Gaspar MJ, Romero E, Lara C, Santander C, Torrealba L, Savescu T, Hermida C. Phase IV noninferiority controlled randomized trial to evaluate the impact on diagnostic thinking and patient management and the test-retest reproducibility of the Gaxilose test for hypolactasia diagnosis. Medicine (Baltimore). 2018 Nov;97(46):e13136. doi: 10.1097/MD.0000000000013136. PMID 30431582